CLINICAL TRIAL: NCT02431403
Title: Open-labeled, Multicenter, Phase I/II Study of Imatinib Combined With ESHAP as Salvage Therapy in Relapsed/Refractory Non-Hodgkin's Lymphoma
Brief Title: ESHAP-Imatinib for Refractory/Relapsed Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jooseop Chung, Professor department of hematooncology, Pusan National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMACEL
Record Dates: First submitted 2015-04-21; First posted 2015-05-01 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ESHAP-Imatinib 100mg (Experimental): Imatinib 100 mg combined with ESHAP
  * ESAHP D1-4 Etoposide 40mg/m2 D1-4 Cisplatin 25mg/m2 D5 Cytarabine 2000mg/m2 D1-5 Methylprednisolone 250mg/m2 D6 Pegfilgrastim 6mg
  Interventions: Drug: ESHAP-Imatinib
- ESHAP-Imatinib 200mg (Experimental): Imatinib 200 mg combined with ESHAP
  * ESAHP D1-4 Etoposide 40mg/m2 D1-4 Cisplatin 25mg/m2 D5 Cytarabine 2000mg/m2 D1-5 Methylprednisolone 250mg/m2 D6 Pegfilgrastim 6mg
  Interventions: Drug: ESHAP-Imatinib
- ESHAP-Imatinib 400mg (Experimental): Imatinib 400 mg combined with ESHAP
  * ESAHP D1-4 Etoposide 40mg/m2 D1-4 Cisplatin 25mg/m2 D5 Cytarabine 2000mg/m2 D1-5 Methylprednisolone 250mg/m2 D6 Pegfilgrastim 6mg
  Interventions: Drug: ESHAP-Imatinib
- ESHAP-Imatinib 300mg (Experimental): Imatinib 300 mg combined with ESHAP
  * ESAHP D1-4 Etoposide 40mg/m2 D1-4 Cisplatin 25mg/m2 D5 Cytarabine 2000mg/m2 D1-5 Methylprednisolone 250mg/m2 D6 Pegfilgrastim 6mg
  Interventions: Drug: ESHAP-Imatinib

INTERVENTIONS:
Drug: ESHAP-Imatinib — After selection of the maximum-tolerated dose of the combination ESHAP with imatinib a phase 2 of the study will be performed in order to evaluate the ORR of ESHAP-imatinib.

SUMMARY:
Open-labeled, multicenter, phase I/II study of imatinib combined with ESHAP as salvage therapy in relapsed/refractory non-Hodgkin's lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed non-Hodgkin's lymphoma, refractory or relapsed after 1st line treatment.
2. Paraffin block of the lesions available for immunohistochemical analysis
3. Candidate for ESHAP salvage therapy
4. Evidence of at least one lesion with a diameter of 1.5 cm
5. Age of over 20 years
6. Eastern cooperative oncology group performance status (ECOG) less than or equal to 2.
7. Adequate kidney function with serum creatinine< 2.5 mg/dL, creatinine clearance ≥ 50 mL/min
8. Adequate liver function with aspartate transaminase (AST)/alanine aminotransferase (ALT) lower than or equal to 3 times the normal upper limit; Total bilirubin lower than or equal to 1.5 times the upper limit ;alkaline phosphatase lower than or equal to 5 times the normal upper limit.
9. Adequate bone marrow function with absolute neutrophil count ≥ 1,000/uL; platelets ≥ 75,000/uL; hemoglobin ≥ 9.0 g/dL
10. Patients who gave voluntarily informed consent before performing any test test that is not part of routine care of patients

Exclusion Criteria:

1. Patients with history of exposure to imatinib or other Bcr-Abl tyrosine-kinase inhibitors
2. Known or suspected hypersensitivity to imatinib
3. Potential use or usage alteration of CYP3A4 inducers or inhibitors from prior to 21 days of to the test regimen until the initiation of round 2 ESHAP. Exceptions are itraconazole and fluconazole for treatment or prevention of fungal infection, hydrocortisone and dexamethasone for treatment of nausea/vomiting/fluid retention, and methylprednisolone as a part of the ESHAP regimen.
4. Known involvement of the central nervous system (CNS) by lymphoma.
5. Pregnant or breast-feeding. Females of childbearing potential who do not agree to undergo pregnancy tests or repeated use effective birth control while included in the clinical trial.
6. Serious or uncontrolled medical condition, such as presence of abnormal or clinically significant cardiac disease, such as acute myocardial infarction or unstable angina within 6 months prior to initiation of treatment with ESHAP-imatinib, serious neurological or psychological conditions such as dementia or epilepsy, or uncontrolled active infection.
7. Prior history of malignancy other than to non-Hodgkin's lymphoma (except basal or squamous cell skin and in situ carcinoma of the cervix) unless the patient free of disease beyond 5 years are.
8. HIV positive and in treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2015-02; Primary Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | Up to 33 weeks
  Adverse events are recorded and analyzed from the time of enrollment to last day of ESHAP-imatinib treatment

SECONDARY OUTCOMES:
Phase I/II Overall Response Rate (ORR) | Week 4, Week 10, Week 16
Phase II Event-Free Survival | Up to 3 years
Phase II Overall Survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jooseop Chung, Principal Investigator — Pusan National Universty Hospital
Locations (5):
- South Korea (5):
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Background] Edling CE, Hallberg B. c-Kit--a hematopoietic cell essential receptor tyrosine kinase. Int J Biochem Cell Biol. 2007;39(11):1995-8. doi: 10.1016/j.biocel.2006.12.005. Epub 2007 Jan 20. PMID 17350321
- [Background] Escribano L, Ocqueteau M, Almeida J, Orfao A, San Miguel JF. Expression of the c-kit (CD117) molecule in normal and malignant hematopoiesis. Leuk Lymphoma. 1998 Aug;30(5-6):459-66. doi: 10.3109/10428199809057558. PMID 9711908
- [Background] Ikeda H, Kanakura Y, Tamaki T, Kuriu A, Kitayama H, Ishikawa J, Kanayama Y, Yonezawa T, Tarui S, Griffin JD. Expression and functional role of the proto-oncogene c-kit in acute myeloblastic leukemia cells. Blood. 1991 Dec 1;78(11):2962-8. PMID 1720040
- [Background] Pinto A, Gloghini A, Gattei V, Aldinucci D, Zagonel V, Carbone A. Expression of the c-kit receptor in human lymphomas is restricted to Hodgkin's disease and CD30+ anaplastic large cell lymphomas. Blood. 1994 Feb 1;83(3):785-92. PMID 7507733
- [Background] Hongyo T, Li T, Syaifudin M, Baskar R, Ikeda H, Kanakura Y, Aozasa K, Nomura T. Specific c-kit mutations in sinonasal natural killer/T-cell lymphoma in China and Japan. Cancer Res. 2000 May 1;60(9):2345-7. PMID 10811105
- [Background] Melnyk A, Rodriguez A, Pugh WC, Cabannillas F. Evaluation of the Revised European-American Lymphoma classification confirms the clinical relevance of immunophenotype in 560 cases of aggressive non-Hodgkin's lymphoma. Blood. 1997 Jun 15;89(12):4514-20. PMID 9192775
- [Background] Aozasa K, Zaki MA. Epidemiology and pathogenesis of nasal NK/T-cell lymphoma: a mini-review. ScientificWorldJournal. 2011 Feb 14;11:422-8. doi: 10.1100/tsw.2011.41. PMID 21336457
- [Background] Brauns TC, Schultewolter T, Dissemond J, Maschke J, Goos M. C-KIT expression in primary cutaneous T-cell lymphomas. J Cutan Pathol. 2004 Oct;31(9):577-82. doi: 10.1111/j.0303-6987.2004.00182.x. PMID 15330987
- [Background] Choe YS, Kim JG, Sohn SK, Kim DH, Baek JH, Lee KB, Do YR, Kwon KY, Song HS, Lee MH, Park TI. c-kit Expression and mutations in peripheral T cell lymphomas, except for extra-nodal NK/T cell lymphomas. Leuk Lymphoma. 2006 Feb;47(2):267-70. doi: 10.1080/10428190500281680. PMID 16321856
- [Background] Giantin M, Aresu L, Arico A, Gelain ME, Riondato F, Comazzi S, Dacasto M. Evaluation of tyrosine-kinase receptor c-kit mutations, mRNA and protein expression in canine lymphoma: might c-kit represent a therapeutic target? Vet Immunol Immunopathol. 2013 Aug 15;154(3-4):153-9. doi: 10.1016/j.vetimm.2013.05.014. Epub 2013 May 30. PMID 23791075
- [Background] Andrae J, Gallini R, Betsholtz C. Role of platelet-derived growth factors in physiology and medicine. Genes Dev. 2008 May 15;22(10):1276-312. doi: 10.1101/gad.1653708. PMID 18483217
- [Background] Piccaluga PP, Agostinelli C, Califano A, Rossi M, Basso K, Zupo S, Went P, Klein U, Zinzani PL, Baccarani M, Dalla Favera R, Pileri SA. Gene expression analysis of peripheral T cell lymphoma, unspecified, reveals distinct profiles and new potential therapeutic targets. J Clin Invest. 2007 Mar;117(3):823-34. doi: 10.1172/JCI26833. Epub 2007 Feb 15. PMID 17304354
- [Background] Huang Y, de Reynies A, de Leval L, Ghazi B, Martin-Garcia N, Travert M, Bosq J, Briere J, Petit B, Thomas E, Coppo P, Marafioti T, Emile JF, Delfau-Larue MH, Schmitt C, Gaulard P. Gene expression profiling identifies emerging oncogenic pathways operating in extranodal NK/T-cell lymphoma, nasal type. Blood. 2010 Feb 11;115(6):1226-37. doi: 10.1182/blood-2009-05-221275. Epub 2009 Nov 30. PMID 19965620
- [Background] Chen YP, Chang KC, Su WC, Chen TY. The expression and prognostic significance of platelet-derived growth factor receptor alpha in mature T- and natural killer-cell lymphomas. Ann Hematol. 2008 Dec;87(12):985-90. doi: 10.1007/s00277-008-0539-z. Epub 2008 Jul 17. PMID 18633616
- [Background] Passam FH, Alexandrakis MG, Kafousi M, Fotinou M, Darivianaki K, Tsirakis G, Roussou PA, Stathopoulos EN, Siafakas NM. Histological expression of angiogenic factors: VEGF, PDGFRalpha, and HIF-1alpha in Hodgkin lymphoma. Pathol Res Pract. 2009;205(1):11-20. doi: 10.1016/j.prp.2008.07.007. Epub 2008 Oct 23. PMID 18950958
- [Background] Renne C, Willenbrock K, Kuppers R, Hansmann ML, Brauninger A. Autocrine- and paracrine-activated receptor tyrosine kinases in classic Hodgkin lymphoma. Blood. 2005 May 15;105(10):4051-9. doi: 10.1182/blood-2004-10-4008. Epub 2005 Jan 27. PMID 15677564
- [Background] Capdeville R, Buchdunger E, Zimmermann J, Matter A. Glivec (STI571, imatinib), a rationally developed, targeted anticancer drug. Nat Rev Drug Discov. 2002 Jul;1(7):493-502. doi: 10.1038/nrd839. PMID 12120256
- [Background] Ruan J, Luo M, Wang C, Fan L, Yang SN, Cardenas M, Geng H, Leonard JP, Melnick A, Cerchietti L, Hajjar KA. Imatinib disrupts lymphoma angiogenesis by targeting vascular pericytes. Blood. 2013 Jun 27;121(26):5192-202. doi: 10.1182/blood-2013-03-490763. Epub 2013 Apr 30. PMID 23632889
- [Background] Aloyz R, Grzywacz K, Xu ZY, Loignon M, Alaoui-Jamali MA, Panasci L. Imatinib sensitizes CLL lymphocytes to chlorambucil. Leukemia. 2004 Mar;18(3):409-14. doi: 10.1038/sj.leu.2403247. PMID 14712290
- [Background] Shimizu H, Popova M, Fleury F, Kobayashi M, Hayashi N, Sakane I, Kurumizaka H, Venkitaraman AR, Takahashi M, Yamamoto K. c-ABL tyrosine kinase stabilizes RAD51 chromatin association. Biochem Biophys Res Commun. 2009 May 1;382(2):286-91. doi: 10.1016/j.bbrc.2009.03.020. Epub 2009 Mar 11. PMID 19285032
- [Background] Hebb J, Assouline S, Rousseau C, Desjardins P, Caplan S, Egorin MJ, Amrein L, Aloyz R, Panasci L. A phase I study of imatinib mesylate in combination with chlorambucil in previously treated chronic lymphocytic leukemia patients. Cancer Chemother Pharmacol. 2011 Sep;68(3):643-51. doi: 10.1007/s00280-010-1530-7. Epub 2010 Dec 1. PMID 21120481
- [Background] Arefi M, Garcia JL, Briz MM, de Arriba F, Rodriguez JN, Martin-Nunez G, Martinez J, Lopez J, Suarez JG, Moreno MJ, Merino MA, Gutierrez NC, Hernandez-Rivas JM. Response to imatinib mesylate in patients with hypereosinophilic syndrome. Int J Hematol. 2012 Sep;96(3):320-6. doi: 10.1007/s12185-012-1141-7. Epub 2012 Jul 18. PMID 22806436
- [Background] Hollmann CA, Tzankov A, Martinez-Marignac VL, Baker K, Grygorczyk C, Grygorczyk R, Foulkes W, Nadeau J, Dirnhofer S, Aloyz R. Therapeutic implications of Src independent calcium mobilization in diffuse large B-cell lymphoma. Leuk Res. 2010 May;34(5):585-93. doi: 10.1016/j.leukres.2009.08.030. Epub 2009 Sep 16. PMID 19758698
- [Background] Velasquez WS, Cabanillas F, Salvador P, McLaughlin P, Fridrik M, Tucker S, Jagannath S, Hagemeister FB, Redman JR, Swan F, et al. Effective salvage therapy for lymphoma with cisplatin in combination with high-dose Ara-C and dexamethasone (DHAP). Blood. 1988 Jan;71(1):117-22. PMID 3334893
- [Background] Velasquez WS, McLaughlin P, Tucker S, Hagemeister FB, Swan F, Rodriguez MA, Romaguera J, Rubenstein E, Cabanillas F. ESHAP--an effective chemotherapy regimen in refractory and relapsing lymphoma: a 4-year follow-up study. J Clin Oncol. 1994 Jun;12(6):1169-76. doi: 10.1200/JCO.1994.12.6.1169. PMID 8201379
- [Background] Rodriguez MA, Cabanillas FC, Hagemeister FB, McLaughlin P, Romaguera JE, Swan F, Velasquez W. A phase II trial of mesna/ifosfamide, mitoxantrone and etoposide for refractory lymphomas. Ann Oncol. 1995 Jul;6(6):609-11. doi: 10.1093/oxfordjournals.annonc.a059252. PMID 8573542
- [Background] Gutierrez M, Chabner BA, Pearson D, Steinberg SM, Jaffe ES, Cheson BD, Fojo A, Wilson WH. Role of a doxorubicin-containing regimen in relapsed and resistant lymphomas: an 8-year follow-up study of EPOCH. J Clin Oncol. 2000 Nov 1;18(21):3633-42. doi: 10.1200/JCO.2000.18.21.3633. PMID 11054436
- [Background] Zhu Y, Qian SX. Clinical efficacy and safety of imatinib in the management of Ph(+) chronic myeloid or acute lymphoblastic leukemia in Chinese patients. Onco Targets Ther. 2014 Mar 6;7:395-404. doi: 10.2147/OTT.S38846. eCollection 2014. PMID 24623982
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396